CLINICAL TRIAL: NCT01068574
Title: Evaluation of the BASIC Scale (Basic Assessment of Severity of Illness in Children): A Simple Triage Tool for Resource-limited Settings
Brief Title: Evaluation of the Basic Assessment of Severity of Illness in Children (BASIC) Scale
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Partners in Health (Other); Thrasher Research Fund (Other); Ministry of Health, Rwanda (Other Government)
Responsible Party: Peter Drobac, MD, Brigham and Women's Hospital
Other Study IDs: 2009P002546
Record Dates: First submitted 2010-02-12; First posted 2010-02-15 (Estimated); Last update posted 2010-08-03 (Estimated); Status verified 2010-08

CONDITIONS: Acute Illness
Keywords: Acute illnesses in children under five

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Single Observational Cohort
  Interventions: Other: BASIC Score (Observational)

INTERVENTIONS:
Other: BASIC Score (Observational) — The BASIC Score will be assessed by a study staff, but there are no interventions.

SUMMARY:
The purpose of this study is to assess whether the BASIC Scale--a simple, non-invasive clinical triage protocol--predicts severe illness, hospitalization or death among children under age five presenting for acute care in a rural African health center.

ELIGIBILITY:
Inclusion Criteria:

* Child aged two months to five years presenting routine or urgent care in an ambulatory facility

Exclusion Criteria:

* None

Ages: 2 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged two months to five years presenting to a rural health center in Rwanda.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-09 (Estimated); Study Completion 2010-09 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Butaro Health Centre, Butaro, Northern Province, Rwanda